CLINICAL TRIAL: NCT03347318
Title: Non-interventional Study for the Determination of Molecular Resistance Profiling to Targeted Therapies in Patients With Neoplastic Disease
Brief Title: Target Therapies Resistance Molecular Profiling in Patients With Neoplastic Disease
Acronym: PROFILING
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Other Study IDs: 001-IRCC-00IIS-10
Record Dates: First submitted 2017-07-18; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-07

CONDITIONS: Solid Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, saliva, feces, urine and tumor specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main purpose of this study is to define the molecular profile of selected solid tumors. From each participants will be collected biological materials for molecular analysis, including saliva, blood and vital tumor tissue derived form surgical or biopsy procedures. Whereas possible, vital tumor specimens will be inoculated and propagated in immunocompromised NOD/SCID mice to study the genetic correlations between genetic status and response to target drugs.

ELIGIBILITY:
Inclusion Criteria:

Patients with at least one of the following selected solid tumors:

* Colorectal Cancer (primary or with synchronous/metachronous liver metastases)
* Prostate Cancer
* Head & Neck Tumors
* Gastric Cancer
* Glioblastoma
* Breast Cancer
* Hepatocarcinoma
* Biliary Tract Carcinoma
* Lung Cancer (primary)
* Rare Tumors (incidence ≤ 5x10-6)
* Metastatic Sarcoma
* Metastatic Melanoma

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with selected solid tumors (CRC, Prostate Cancer, Head & Neck Cancer, Gastric Cancer, Glioblastoma, Breast Cancer, Hepatocarcinoma, Biliary Tract Carcinoma, Lung Cancer, Rare Tumors, Metastatic Sarcoma and Metastatic Melanoma).
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2011-01; Primary Completion 2018-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
number of patient correctly sampled | through study completion, an average of five years
  number of patients with biological samples idoneous for molecular profiling testing (nucleic acid extraction, protein) over all recruited patients.

SECONDARY OUTCOMES:
number of patients with detected genetic alterations that respond to treatments assigned by physician. | through study completion, an average of five years

CONTACTS AND LOCATIONS:
Locations (15):
- Italy (15):
  - Ospedale Regionale Umberto Parini, Aosta
  - Policlinico S.Orsola Malpighi, Bologna
  - Istituto Di Candiolo - Fondazione Del Piemonte Per L'Oncologia (FPO-Irccs), Candiolo
  - Azienda Ospedaliero-Universitaria Careggi, Genova
  - Azienda Ospedaliera Niguarda Ca'Granda, Milan
  - IEO - Istiuto Europeo di Oncologia, Milan
  - Fondazione IRCCS - Istituto Nazionale dei Tumori, Milan
  - AOU S. Luigi Gonzaga, Orbassano
  - IOV - Istituto Oncologico Veneto, Padua
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Policlinico Universitario Campus Biomedico, Roma
  - A.O. Città della Salute e della Scienza di Torino - Presidio ospedaliero Ostetrico Ginecologico Sant'Anna, Turin
  - AOU Città della Salute e della Scienza di Torino - Presidio Molinette, Turin
  - Ospedale Mauriziano Umberto I, Turin
  - Presidio Ospedaliero Martini, Turin